CLINICAL TRIAL: NCT02518919
Title: Procedural Sedation And Analgesia in Children in the Emergency Department: The Role of Adjunct Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Michigan (Other)
Responsible Party: Principal Investigator, Nirupama Kannikeswaran, Associate Professor of Pediatrics and Emergency Medicine, Children's Hospital of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R1-2014-79
Record Dates: First submitted 2015-08-03; First posted 2015-08-10 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Conscious Sedation
Keywords: Children; Emergency Department; Sedation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard (No Intervention): Patients will receive intravenous ketamine (1-2mg/kg)
- Child Life Intervention (Experimental): Child life therapist will comfort the child during all painful procedures(including IV insertion) and during sedation
  Interventions: Other: Child life intervention
- Music Listening (Experimental): Patients will listen to music of their choice using headphones during sedation
  Interventions: Other: Music listening

INTERVENTIONS:
Other: Child life intervention — The participants will receive IV ketamine for sedation. In addition in this arm, 'Child Life Intervention', comfort measures provided by a trained child life therapist during painful procedures.
  Arms: Child Life Intervention
Other: Music listening — The participants will receive IV ketamine for sedation. In addition in this arm, 'Music Listening' to music chosen by the patient using headphones
  Arms: Music Listening

SUMMARY:
The role of Adjunct therapies such as Child Life therapy and Music listening during Procedural Sedation and Analgesia(PSA) for children during painful procedures has not been studied in the Emergency Department (ED). The investigators hypothesize that there will be a reduction in sedation medication dosage without change in sedation efficacy by addition of music therapy and Child Life to standard sedation protocol in children 3-15 years of age who undergo PSA for painful (orthopedic procedures, laceration repair, incision and drainage) procedures in a Pediatric emergency Department (PED).

DETAILED DESCRIPTION:
The investigators propose to perform a prospective randomized control trial on children aged 3-15 years of age who undergo PSA for painful procedures (orthopedic procedures, laceration repair, incision and drainage of abscess) at Children's Hospital of Michigan Emergency Department. The investigators will study the effect of child life specialist intervention and listening to music on the sedation medication requirement and sedation efficacy in those patients undergoing orthopedic procedures under PSA with intravenous ketamine Patients will be randomly allocated to one of the three groups: 1) Standard sedation protocol 2) standard sedation protocol with listening to music and 3) standard sedation protocol with child life intervention. This will be done by opening the double sealed envelope after obtaining informed consent from the parents/legal guardians. In addition, an assent will also be obtained from all children older than 7 years of age.

Study Intervention: Study population will be divided into 3 groups: 1) Standard sedation protocol 2) Standard sedation protocol with child life intervention and 3) Standard sedation protocol with music listening. All children enrolled in this study will receive sedation only after a pre sedation assessment has been performed using current institutional guidelines as has been applied to all ED sedation patients. Participants will be monitored using published sedation guidelines with measurements of vital signs, pulse oximetry at baseline, every 5 minutes during the procedure and post procedure for the entire duration of sedation. The dose of sedation medication administered will be at the discretion of the sedation physician and the study research assistant will not participate in any of the clinical procedures. For those participants assigned to the child life intervention group, trained child life personnel will introduce the procedure to the child and the family and will provide comforting measures appropriate to the age of the patient during the placement of intravenous line and throughout the procedure. The participants assigned to the music therapy group will be asked to choose a music of their choice which they will listen via head phones.

The investigators will collect the following variables: patient demographics, American Society of Anesthesiologists classification, indication for the sedation, sedation medication dosage, need for re-dosing, sedation related adverse events and ED disposition. In addition specifically for this study, the investigators will assess the pre-sedation agitation ,sedation efficacy using Ramsey Sedation Scale, pain scale using FACES-P and parent and consultant satisfaction using a 3-point Likert scale(very satisfied, satisfied, not satisfied). The Ramsey Sedation Scoring and FACES-P scoring will be performed by a trained research assistant who will be blinded to the sedation medication dosage at the following three time periods: just prior to administration of ketamine, during sedation and during recovery just prior to patient discharge.

In addition, the study research assistant will also complete a follow-up phone call within 72 hours after discharge from the ED to the parents/guardians of the children to evaluate for the particpant's experience with the sedation(the pain they perceived during the procedure, their memory of the event) and adverse events that occur at home.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-15 years
* American Society of Anesthesiologists (ASA) classification 1 or 2
* Receiving intravenous ketamine for PSA for painful procedures such as fracture/joint reduction, laceration repair, incision drainage of abscess .

Exclusion Criteria:

1. Known contraindications, allergy or previous adverse events with ketamine
2. Receive intramuscular or oral sedation or sedation medications other than ketamine
3. Receive ketamine for procedures not listed above
4. Outside the age range listed above
5. Parents/guardians refuse study participation.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2016-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Michigan, Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Lepage C, Drolet P, Girard M, Grenier Y, DeGagne R. Music decreases sedative requirements during spinal anesthesia. Anesth Analg. 2001 Oct;93(4):912-6. doi: 10.1097/00000539-200110000-00022. PMID 11574356
- [Background] Koch ME, Kain ZN, Ayoub C, Rosenbaum SH. The sedative and analgesic sparing effect of music. Anesthesiology. 1998 Aug;89(2):300-6. doi: 10.1097/00000542-199808000-00005. PMID 9710387

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were screened for eligibility using electronic medical records and if eligible were approached by the study Research Assistant(RA) for informed consent. If the parent/guardian refused participation, were non- English speaking and if parent/legal guardian was not present to complete the informed consent process they were excluded from study
Period: Overall Study
Arm/Group | Standard | Music Listening | Child Life Intervention
Started | 21 | 21 | 21
Completed | 20 | 20 | 19
Not Completed | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | Music Listening | Child Life Intervention | Total
Number analyzed (Participants) | 20 | 20 | 19 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5 [4.5 to 9.5] | 8.5 [6.5 to 11] | 9 [6 to 11] | 8 [5 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 13 | 27
  Male | 12 | 14 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 18 | 20 | 17 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 3 | 6
  Caucasian | 4 | 9 | 3 | 16
  African American | 12 | 9 | 10 | 31
  Mixed | 0 | 1 | 0 | 1
  Others | 2 | 0 | 3 | 5
American Society of Anesthesiologists(ASA) Classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists physical status classification is a system to assess fitness prior to surgery/procedure.
  ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation The addition of "E" denotes Emergency surgery Higher the ASA class higher the risk from sedation and procedure
  Participants
    American Society of Anesthesiologist, ASA I | 16 | 15 | 16 | 47
    American Society of Anesethesiologist, ASA II | 4 | 5 | 3 | 12
Procedure Type [Count of Participants; unit: Participants]
  fracture/dislocation reduction | 12 | 16 | 13 | 41
  Incision and drainage | 1 | 1 | 2 | 4
  laceration repair | 7 | 3 | 4 | 14
Pre - sedation pain medication [Count of Participants; unit: Participants]
  Pre sedation pain medication yes | 14 | 10 | 14 | 38
  Pre sedation pain medication no | 6 | 10 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Sedation Medication Requirement
Description: Total mg/kg of sedation medication administered IV
Time Frame: Right at the end of the procedure
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Standard | Music Listening | Child Life Intervention
Number analyzed (Participants) | 20 | 20 | 19
mg/kg | 1.58 (0.44) | 1.68 (0.36) | 1.42 (0.47)

2. Secondary Outcome: Sedation Efficacy
Description: compare sedation efficacy among the 3 groups using Ramsey sedation scales and FACES -P (FACES-Pediatric)scale. The Ramsey sedation scales scores sedation at six different levels, according to how arousable the patient is. The continuum of sedation is measured from 1-6 with higher values representing a deeper level of sedation.
  1. Patient is anxious and agitated or restless, or both
  2. Patient is co-operative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response The Faces- PScale is a self-report measure used to assess the intensity of children's pain. The scale ranges from 0 to 10 with 0 indicating no hurt or discomfort to 10 :hurts most/worst
Time Frame: During the Procedure
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Standard | Music Listening | Child Life Intervention
Number analyzed (Participants) | 20 | 20 | 19
scores on a scale
  Ramsay Sedation Score during sedation | 6 [4 to 6] | 6 [4 to 6] | 6 [5 to 6]
  FACES-Pediatric during sedation | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Adverse Events
Description: describe the adverse events experienced by study participants secondary to sedation medication and interventions performed to overcome them
Time Frame: during procedure until discharge from the Emergency Department
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Music Listening | Child Life Intervention
Number analyzed (Participants) | 20 | 20 | 19
Participants | 4 | 8 | 5

4. Secondary Outcome: Number of Participants With Consultant Satisfaction Rating as Either" Not Satisfied", "Satisfied", or "Very Satisfied,"
Description: Compare consultant satisfaction among three groups using Likert scale
Time Frame: within two hours of completion of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Music Listening | Child Life Intervention
Number analyzed (Participants) | 20 | 20 | 19
Participants
  Not satisfied | 0 | 0 | 0
  Satisfied | 13 | 8 | 6
  Very Satisfied | 7 | 12 | 13

5. Secondary Outcome: Number of Participants Who Were re- Dosed With Sedation Medication
Description: compare the need for additional dosages of sedation medication among three groups
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Music Listening | Child Life Intervention
Number analyzed (Participants) | 20 | 20 | 19
Participants | 9 | 4 | 8

ADVERSE EVENTS:
Arm/Group | Standard | Music Listening | Child Life Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 4/20 | 8/20 | 5/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard (N=20) | Music Listening (N=20) | Child Life Intervention (N=19)
Oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) — Oxygen saturation of <90%
Emesis (Gastrointestinal disorders) | 3 (3) | 8 (8) | 3 (3) — Vomiting

LIMITATIONS AND CAVEATS:
Study was a convenience sample. Small sample size. Study could not be blinded for obvious reasons. We did not study active music therapy but evaluated only music listening. We did not control for type of procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No